CLINICAL TRIAL: NCT07340931
Title: Pilot Study on the Adaptation and Tolerance of Essilor® Myopia-control Spectacle Lenses
Acronym: STELLAR
Status: Not yet recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: AP_PL_Stellar
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Myopia
Keywords: myopia; visual correction; compliance
MeSH Terms: conditions — Myopia; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pediatric patient with Essilor® myopia-control spectacle lenses: pediatric patient with Essilor® myopia-control spectacle lenses Stellet 2.0

SUMMARY:
This observational pilot study aims to evaluate the adaptation and tolerance of Essilor® Stellest® myopia-control spectacle lenses in children with progressive myopia. The objective is to assess real-life compliance and comfort during lens wear, as these factors are essential for long-term therapeutic adherence and overall visual health outcomes

DETAILED DESCRIPTION:
Myopia is a refractive error in which light rays from distant objects focus in front of the retina, resulting in blurred distance vision. It is most commonly caused by an elongation of the axial length of the eye. Myopia has become a major public health issue of the 21st century, with estimates suggesting that nearly 50% of the global population will be myopic by 2050. High myopia significantly increases the risk of serious ocular complications, including glaucoma, early cataract, myopic maculopathy, retinal tears, and detachments. Myopia typically begins in childhood and tends to appear earlier and progress faster than in previous generations, with onset now occurring around 6-7 years of age instead of 12-13. Early detection and appropriate optical correction can have a substantial impact on a child's academic performance and quality of life, as good vision is closely linked to both. Progressive myopia, a form that worsens over time, requires active management to slow or halt its progression and prevent high myopia. Among available approaches, optical devices such as Essilor® Stellest® lenses have shown promise in myopia control. However, their real-world effectiveness depends not only on optical performance but also on the child's ability to adapt to and tolerate the lenses, which directly influences daily wear time and long-term compliance. This observational study therefore focuses on evaluating the adaptation and tolerance of Essilor® Stellest® lenses prescribed to children with progressive myopia in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 6 to 16 years with progressive myopia.

Spherical equivalent ≤ -0.50 D under cycloplegia and presence of at least one risk factor (age < 10 years, progression ≥ 0.50 D/year, axial length increase ≥ 0.2 mm/year, high myopia ≤ -6.00 D and/or axial length ≥ 26 mm, both parents myopic, at least one parent highly myopic, or Asian origin).

Patient covered by the French social security system.

Patient and legal guardians providing oral non-opposition to participate in the study.

Exclusion Criteria:

* Patients with strabismus, amblyopia, or syndromic myopia

Ages: 6 Years to 16 Years | Sex: All
Age Groups: Child
Study Population: Children and adolescents with myopia followed at the Ophthalmology Departments of Nantes University Hospital and Strasbourg University Hospital, as well as at the Centre Ophtalmologique de l'Hippodrome in Lambersart.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Adaptation and tolerance of Essilor® Stellest® 2.0 myopia-control spectacle lenses | At 6 months after initiation of lens wear
  Evaluation of the adaptation and tolerance of Essilor® Stellest® 2.0 lenses in children with progressive myopia, using the PREP-2 quality-of-life questionnaire (56 items) to assess comfort, visual satisfaction, and overall acceptance after regular use.